CLINICAL TRIAL: NCT05844397
Title: Comparison of Clinical Outcomes of SMILE vs. LASIK Using Contoura With Phorcides
Brief Title: SMILE vs. LASIK Using Contoura With Phorcides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2023.052
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-03

CONDITIONS: Myopia; Astigmatism
Keywords: SMILE; LASIK; Countoura; Phorcides
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective randomized contralateral study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LASIK using Contoura with Phorcides (Active Comparator): LASIK using Contoura with Phorcides in one eye.
  Interventions: Device: WaveLight EX500 Excimer Laser System
- SMILE (Active Comparator): small incision lenticule extraction (SMILE) refractive surgery on the contralateral eye.
  Interventions: Device: VisuMax Surgical Laser

INTERVENTIONS:
Device: WaveLight EX500 Excimer Laser System — LASIK Refractive Surgery Using Contura with Phorcides
  Arms: LASIK using Contoura with Phorcides
Device: VisuMax Surgical Laser — SMILE Refractive Surgery
  Arms: SMILE

SUMMARY:
Subjects will undergo SMILE surgery in one eye and LASIK using Contoura with Phorcides on the contralateral eye to correct myopia.

DETAILED DESCRIPTION:
Once consented to participate in the study, subjects will have a comprehensive ocular examination to determine eligibility to undergo simultaneous SMILE surgery in one eye and LASIK using Contoura with Phorcides on the contralateral eye to correct myopia.The study objective is to compare the 6-month visual outcomes (i.e., visual acuity, contract sensitivity, high order aberrations), quality of vision (i.e., double vision, glare, starburst, halos, etc.) and dry eye symptoms of patients undergoing contralateral LASIK using Contoura with Phorcides and SMILE surgery. Surgical treatment will be randomized so there is a 50% chance to receive SMILE on the right eye and LASIK on the contralateral eye. Subjects will receive standard of care topical ophthalmic antibiotic and steroid drops. Visual outcomes and patient self-reported symptoms will be assessed at week 2, month 1, month 3, and month 6.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females between the ages of 21 and 50
* Nearsightedness between -2.00 diopters and -8.00 diopters
* Have similar levels of nearsightedness in each eye (≤1.5D of difference between eyes)
* Less than or equal to 3.00 diopters of astigmatism
* Have similar levels of astigmatism in each eye (≤0.75D of difference between eyes)
* Total spherical equivalent (SE) of no more than -8.0 D
* Tricare Prime Beneficiary
* Residing within 60 miles radius from Lackland AFB

Exclusion Criteria:

* Subjects with corneal abnormal findings including signs of keratoconus, keratoconus suspect, abnormal corneal topography, epithelial basement membrane disease, pellucid marginal degeneration, corneal degenerations, progressive and unstable myopia, irregular or unstable corneal mires on central keratometry images, and patients whose corneal thickness would cause anticipated treatment would violate the posterior 250 microns (μm) of corneal stroma from the corneal endothelium.
* Subjects with active collagen vascular, connective tissue, autoimmune or immunodeficiency diseases
* Pregnant or nursing females
* Systemic disease likely to affect wound healing, such as uncontrolled diabetes and severe atopy
* Any ocular disease such as advanced/uncontrolled glaucoma, severe dry eye, active eye infection or inflammation, recent herpes eye infection or problems resulting from past infection.
* 0.25 or 0.50 of manifest astigmatism in either eye
* Taking the medication Isotretinoin (Accutane) or antimetabolites for any medical condition.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Percentage of eyes with Uncorrected Visual Acuity of 20/16 or better at 6-month Post-Op | 6-month Post-Op
  Post-operative uncorrected visual acuity of 20/16 or better measure with ETDRS chart; unit = percentage eyes with Uncorrected Visual Acuity

SECONDARY OUTCOMES:
Change in high contrast visual acuity at 6-month Post-Op | Change from baseline (pre-op) to 6-month Post-Op
  Change in the mean uncorrected visual acuity (unit = logMAR) measure with ETDRS chart from baseline (pre-op) at 6 months post-op.
Change in refractive error at 6-month Post-Op | Change from baseline (pre-op) to 6-month Post-Op
  Change in the mean refractive error measure with phoropter (unit = diopters) from baseline (pre-op) at 6 months post-op.

OTHER OUTCOMES:
Change in low contrast visual acuity at 6-month Post-Op | Change from baseline (pre-op) to 6-month Post-Op
  Change in the mean low contrast visual acuity (unit = logMAR) measure with ETDRS 5% chart from baseline (pre-op) at 6 months post-op.
Change in higher order aberrations at 6-month Post-Op | Changes from baseline (pre-op) to 6-month Post-Op
  Change in the mean higher order aberrations (unit = root mean square) measure with iDesign 2.0 Refractive Studio from baseline (pre-op) at 6 months post-op.
Change in mean score Patient-Reported Outcomes with LASIK Symptoms and Satisfaction (PROWL-SS) Questionnaire at 6-month Post-Op | Changes from baseline (pre-op) to 6-month Post-Op
  The PROWL-SS is a validated tool to assess self-reported symptoms and satisfaction after refractive surgery. Possible Satisfaction Score ranges from 1 (completely satisfied) to 6 (completely dissatisfied). Lower value indicates higher satisfaction. Possible Symptoms Score ranges from 1 (extremely bothersome) to 5 (not at all bothersome). Lower value indicates worse symptoms.
Change in mean score Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire at 6-month Post-Op | Changes from baseline (pre-op) to 6-month Post-Op
  The SPEED is a validated tool to assess self-reported dry eye symptoms. Possible dry eye symptoms score ranges from 0 (never) to 3 (Constant). Higher value indicates worse dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Charisma B Evangelista, MD, Principal Investigator — 59th Medical Wing
Locations (1):
- Joint Warfighter Refractive Surgery Center at WHASC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma KK, Manche EE. Patient-reported quality of vision in a prospective randomized contralateral-eye trial comparing LASIK and small-incision lenticule extraction. J Cataract Refract Surg. 2023 Apr 1;49(4):348-353. doi: 10.1097/j.jcrs.0000000000001127. PMID 36539217